CLINICAL TRIAL: NCT05824962
Title: A Non-invasive Diagnostic Model for Intestinal Fibrosis in Crohn's Disease Based on 18F-FAPI PET Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiao Chen (Other)
Responsible Party: Sponsor-Investigator, Xiao Chen, Director of Nuclear Medicine Department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Other Study IDs: 2022355
Record Dates: First submitted 2023-04-06; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; FDG; FAPI; Fibrosis; PET/CT
MeSH Terms: conditions — Crohn Disease; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — surgical bowel resection specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Crohn's disease (CD) is a chronic transmural inflammatory bowel disease. Prolonged episodes of inflammation can lead to intestinal fibrosis, leading to intestinal stenosis and obstruction. Inflammatory stenosis can be alleviated through anti-inflammatory treatment, while fibrotic stenosis requires endoscopic dilation or surgical treatment. Early detection of the presence and severity of intestinal fibrosis in CD is the key to treatment strategies. Currently, there are certain limitations in the non-invasive evaluation methods for intestinal fibrosis, and it is urgent to develop a new imaging method to achieve non-invasive diagnosis of the degree of fibrosis.

Fibroblast activation protein (FAP) is a marker of intestinal fibrosis in CD. Based on the principle that fibroblast activation protein inhibitor (FAPI) can specifically bind to FAP, FAPI radioactive tracers can achieve targeted tracing and quantification of FAP in vivo. Therefore, 18F-FAPI positron emission tomography (PET) imaging technology has a good application prospect in the noninvasive diagnosis and evaluation of CD intestinal fibrosis.

Based on the successful testing of 18F-FAPI PET imaging in the early stage of the project team to evaluate the nature of CD intestinal stenosis, this project intends to take patients with CD intestinal stenosis as the research object, and use postoperative histopathological analysis as a reference index to evaluate the role of 18F-FAPI combined with 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose(18F-FDG) PET imaging in the qualitative diagnosis of CD intestinal wall fibrosis, as well as the differential diagnosis ability of inflammatory and fibrous stenosis in CD patients, and establish a diagnostic model and evaluation system. Achieving a noninvasive, stable, and objective diagnosis and evaluation of the degree of intestinal fibrosis in CD patients at the molecular level will provide imaging evidence for treatment decision-making, progress, and prognosis of CD patients, and also play an important support role in the development of anti fibrosis drugs, selection of suitable patients, and efficacy evaluation.

DETAILED DESCRIPTION:
This study is a prospective, multicenter study and has been approved by the ethics committee. The subjects of this study were from January 1, 2023 to December 31, 2025.The detailed description is as follows：

1. Patients: The subjects we selected are adults who are not restricted by gender. For details, please refer to the "Eligibility Criteria" column.
2. Clinical data collection: Record the course of disease, PET/computed tomography (CT) examination, computed-tomography enterography(CTE) examination and surgical interval, lesion location, CD activity index, laboratory examination (blood routine, C-reactive protein, erythrocyte sedimentation rate), and other information of all patients.
3. CTE image analysis： Record and evaluate the following indicators: location and length of abnormal small intestine segments, intestinal stenosis, intestinal wall thickness, pre stenosis dilation, ratio of proximal small intestine dilation diameter to the minimum lumen diameter within the stenosis. In addition, record submucosal edema, submucosal fat infiltration, adjacent mesenteric inflammation, abdominal abscess, fistula, etc.
4. PET image analysis: Record and evaluate the following indicators: the maximum, mean and peak standardized uptake value (SUVmax, SUVmean and SUVpeak), Metabolic lesion volume (MLV), total lesion glycolysis (TLG).
5. Pathological analysis: After surgery, the most significant lesion of the intestinal wall was removed for pathological staining. Select normal specimens near the surgical resection edge as the control group. The hematoxylin and eosin (H&E) staining was used to evaluate intestinal wall inflammation; Masson staining was used to evaluate intestinal fibrosis; Immunohistochemical analysis was used to investigate the expression of FAP and glucose transporter protein 1 (GLUT-1).
6. Statistical analysis: Spearman correlation analysis was used to evaluate the correlation between intestinal wall FAP expression level and fibrosis score, as well as the correlation between imaging indicators and fibrosis score, inflammation score, and FAP expression level. Single factor analysis of variance was used to compare the imaging indicators of intestinal wall in four groups with different degrees of fibrosis, and the least significant difference(LSD) method was used for pairwise comparison. Using multivariate logistic regression analysis, and using the forward method and likelihood ratio test to screen variables, independent factors were determined for predicting intestinal fibrosis in lesions using the column chart. Based on the results of multivariate logistic regression analysis, a column chart prediction model was established using the "RMS" program package in R3.6.1 software. The Harrell consistency index of the model construction group was calculated, and a bootstrap calibration curve was drawn to internally verify the predictive performance of the column chart. The Harrell consistency index of the model validation group was calculated to externally verify its predictive performance. Evaluate the diagnostic performance of each variable using subject operated characteristic curve analysis, and calculate the area, sensitivity, specificity, and threshold under each variable curve. Compare the diagnostic efficacy of PET/CT and CTE using Medcalc software.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with CD based on clinical, imaging, endoscopic, and histopathological criteria;
2. Patient age ≥ 18 years old;
3. Within 15 days before surgery, 18F-FAPI, 18F-FDG PET/CT intestinal imaging, and routine CTE imaging were performed;
4. Surgical resection of intestinal segments and imaging evaluation of intestinal segment matching;
5. The pathological analysis of surgical specimens includes H&E, Masson, GLUT1 and FAP immunohistochemical staining;
6. The patient voluntarily participates and signs an informed consent form.

Exclusion Criteria:

1. Pregnant or lactating patients;
2. The quality of imaging images is poor and cannot be used for diagnosis and evaluation;
3. If the pathological section of the specimen does not cover the entire intestinal wall;
4. The fasting blood glucose level is higher than 11.1mmol/L;
5. Patients with contraindications for CTE examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects we selected are adults who are not restricted by gender. For details, please refer to the "Eligibility Criteria" column.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Histologic Scores for Inflammatory | Completed within one week after surgery
  Paraffin section specimens were stained by using hematoxylin and eosin for the histologic inflammation score. Two pathologists graded the histologic slices from the most severe areas for inflammation by using a semiquantitative scoring system. The inflammation score was scored between 0 and 3 points as follows: 0: none (No inflammation or distortion), 1: mild (Lamina propria inflammation only), 2: moderate (Submucosal foci of inflammation and/or foci of transmural inflammation), 3: severe (Significant, dissecting, confluent transmural inflammation).
Histologic Scores for Fibrotic | Completed within one week after surgery
  Paraffin section specimens were stained by using Masson trichrome for the histologic fibrosis score. Two pathologists graded the histologic slices from the most severe areas for fibrosis by using a semiquantitative scoring system. The fibrosis score was scored between 0 and 3 points as follows: 0: none (No fibrosis), 1: mild (Minimal fibrosis in submucosa or subserosa), 2: moderate (Increased submucosal fibrosis, septa into muscularis propria and/or septa through muscularis propria, increase in subserosal collage), 3: severe (Significant transmural scar, marked subserosal collagen).
Metabolic parameters | Completed within one week after PET examination
  Total Lesion Glycolysis (TLG) of bowel lesions are measured on PET.

SECONDARY OUTCOMES:
FAP expression and SUV | through study completion, an average of 1 year
  Correlation between FAP expression and SUV in PET
GLUT-1 expression and SUV | through study completion, an average of 1 year
  Correlation between GLUT-1 expression and SUV in PET
Inflammatory histological score and SUV | through study completion, an average of 1 year
  Correlation between inflammatory histological score and SUV in PET
Fibrotic histological score and SUV | through study completion, an average of 1 year
  Correlation between fibrotic histological score and SUV in PET

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Chen, Ph.D, Principal Investigator — Daping Hospital, Army Medical University
Locations (1):
- Department of Nuclear Medicine, Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scharitzer M, Macher-Beer A, Mang T, Unger LW, Haug A, Reinisch W, Weber M, Nakuz T, Nics L, Hacker M, Bergmann M, Rasul S. Evaluation of Intestinal Fibrosis with 68Ga-FAPI PET/MR Enterography in Crohn Disease. Radiology. 2023 May;307(3):e222389. doi: 10.1148/radiol.222389. Epub 2023 Feb 28. PMID 36853176
- See also: Evaluation of Intestinal Fibrosis with 68Ga-FAPI PET/MR Enterography in Crohn Disease — http://pubmed.ncbi.nlm.nih.gov/33247327/